CLINICAL TRIAL: NCT04252417
Title: Open Label, Phase I Study to Assess and Compare the Pharmacokinetic Parameters After Single Oral Administration of MD1003 100 mg in Hepatic Impaired Patients and Healthy Subjects With Normal Hepatic Function
Brief Title: HI Study to Assess and Compare the Pharmacokinetic Parameters of MD1003 in Hepatic Impaired Patients and Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to other Phase 3 trial failure to meet primary endpoint
Sponsor: MedDay Pharmaceuticals SA (Industry)
Collaborators: Eurofins Optimed (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: MD1003CT201901HI; 2019-002315-26 (EudraCT Number)
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-01

CONDITIONS: Healthy Volunteers; Hepatic Impairment of Moderate Child Pugh Category

STUDY DESIGN:
Intervention Model Description: Open label, Parallel-group, Single oral dose
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with hepatic impaired function (Active Comparator): 8 patients with hepatic impairment of moderate Child Pugh category
  Interventions: Drug: MD1003
- Healthy subjects (Active Comparator): Healthy volunteers will be matched with impaired hepatic function patients
  Interventions: Drug: MD1003

INTERVENTIONS:
Drug: MD1003 — Single oral dose administration of MD1003 at Day 1

SUMMARY:
This is a Phase 1, multicentric, open-label,two arms to assess and compare the effect of single oral administration of MD1003 on the pharmacokinetic parameters in hepatic impaired patients and healthy subjects with normal hepatic function.

The planned enrollment is 16 subjects (8 impaired patients and 8 healthy subjects).

DETAILED DESCRIPTION:
The study is a multicentric, open label, phase I, two arms study to compare pharmacokinetics of MD1003 after a single oral dose of MD1003 100 mg in eight (8) healthy male/female subjects and eight (8) male/female patients of moderate Child Pugh category. Healthy subjects and patients will receive a single oral dose of MD1003 100 mg. The healthy subjects will match with impaired hepatic function patients on ethnic group, sex, age (+/- 10 years) and BMI (+/- 20%).

Participants will be admitted into the Clinical Research Units (CRU) on Day-3. On the morning of Day 1, subjects will receive a single 100 mg oral dose of MD1003 following an overnight fast (i.e., at least 10 hours). Participants will be confined to the CRU until discharge on Day 8, with PK blood sample draws for measurement of MD1003 and its main metabolites being taken throughout the confinement (Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144, 168h post dose). A Follow up post study visit will occur on Day 14 (± 2 days).

Adverse events (AEs), clinical laboratory evaluations, vital signs assessments, 12-lead electrocardiograms (ECGs), and physical examination (PE) findings will be monitored at Screening and at specified times during the study. All AEs will be recorded throughout the study (i.e., from signing of the Informed Consent Form until Study Completion).

The Study Completion is defined as the last subject's end-of-study assessment.

ELIGIBILITY:
Inclusion Criteria:

For eligibility into the trial, subjects and patients must meet all the following inclusion criteria:

1. Male or female subjects, aged 18 to 75 years inclusive;
2. Females participating in this study must be of non-childbearing potential or using acceptable contraception for the full duration of the study and for 1 month after the end of treatment, as described below:

   * Cessation of menses for at least 12 months due to ovarian failure;
   * Surgical sterilization such as bilateral oophorectomy, hysterectomy, or medically documented ovarian failure;
   * Using an acceptable effective non-hormonal method of contraception (bilateral tubal occlusion, vasectomized partner or intra-uterine device, sexual abstinence, male or female condom with spermicide);
3. Negative serum pregnancy test at screening (if applicable);
4. Normal renal function according to the age
5. Non-smoker subject or smoker of not more than 5 cigarettes a day;
6. Signing a written informed consent prior to selection;
7. Covered by Health Insurance System and / or in compliance with the recommendations of National Law in force relating to biomedical research.

For hepatic impaired patients:

1. Hepatic impairment of moderate Child Pugh category determined at screening (Class B: 7 to 9 points);
2. Stable Hepatic dysfunction e.g. no clinical significant change in disease status within the last 30 days documented by recent medical history, including no worsening of clinical signs of hepatic impairment or no worsening of total Bilirubin or Prothrombin time>50%.
3. Stable treatment regimen or dose of medication
4. Supine blood pressure ≤ 170/110 mmHg;
5. Body Mass Index (BMI) between 20 and 34 kg/m² inclusive.

For healthy subject with normal hepatic function:

1. Considered as healthy after a comprehensive clinical assessment (detailed medical history and complete physical examination);
2. Body Mass Index (BMI) between 20 and 30 kg/m2 inclusive and body weight (BW) not lower than 55kg;
3. Normal Blood Pressure (BP) and Heart Rate (HR) at the screening visit after 10 minutes in supine position:

   * 90 mmHg ≤ Systolic Blood Pressure (SBP) ≤ 145 mmHg,
   * 50 mmHg ≤ Diastolic Blood Pressure (DBP) ≤ 90 mmHg,
   * 45 bpm ≤ HR ≤ 90 bpm,
   * Or considered NCs by investigators;
4. Normal ECG recording on a 12-lead ECG at the screening visit:

   * 120 < PR < 220 ms,
   * QRS < 110 ms,
   * QTcf ≤ 430 ms for male and < 450 ms for female,
   * No sign of any trouble of sinusal automatism,
   * Or considered NCs by investigators;
5. Laboratory parameters within the normal range of the laboratory (hematological, blood chemistry tests, urinalysis). Individual values out of the normal range can be accepted if judged clinically non relevant by the Investigator. In particular, the hepatic function should be considered as normal;
6. Normal dietary habits;
7. Matched to at least 1 hepatic impaired patient by ethnic group, sex, age (+/- 10 years) and BMI (+/- 20%).

Exclusion Criteria:

Subjects or Patients meeting any of the following criteria will not be included into the trial:

1. Positive Hepatitis B surface (HBs) antigen or anti Hepatitis C Virus (HCV) antibody, or positive results for Human Immunodeficiency Virus (HIV) 1 or 2 tests);
2. Subject/Patient who, in the judgment of the Investigator, is likely to be non-compliant or uncooperative during the study, or unable to cooperate because of a language problem, poor mental development;
3. Subject/Patient who cannot be contacted in case of emergency;
4. History or presence of allergy or unusual reactions to some drugs or anesthetics or known hypersensitivity to the investigation product or its excipients (including lactose);
5. Any medications intake within 3 months that may interfere with absorption, distribution, metabolism or excretion of the study drug, or any medication that may result in induction or inhibition of microsomal enzymes;
6. Subject/Patient who is in the exclusion period of a previous study;
7. Administrative or legal supervision;
8. Blood donation (including in the frame of a clinical trial) within 2 months before administration or blood donation planned during the study or within 2 months following participation to the study;
9. Subjects/Patients who are pregnant or breastfeeding. Subjects/Patients should not be enrolled if they plan to become pregnant during the time of study participation;
10. Excessive consumption of beverages with xanthine bases (> 4 cups or glasses / day);
11. History or presence of drug abuse;
12. Positive results of screening for drugs of abuse;
13. Intake of any food or any beverage containing grapefruit or grapefruit juice within 48h prior to the first dosing and the inability to stop such intake during the study.
14. Evidence or history of clinically significant hematological, endocrine, pulmonary, gastrointestinal, cardiovascular, renal, psychiatric, neurologic, metabolic, systemic, infectious, or allergic disease (including drug hypersensitivity or allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing);
15. General anesthesia within 3 months before administration;
16. Major surgery within 28 days prior to inclusionor major surgery planned during the next 6 months.

For hepatic impaired patients:

1. Other underlying diseases that may alter Child Pugh components like metastatic cancer to the brain or peritoneal surface or cancer cachexia (hypoalbuminemia, encephalopathy, ascites);
2. History of liver transplant;
3. The patient has an acute exacerbation or unstable hepatic function, as indicated by worsening of clinical and/or laboratory signs of hepatic impairment, within the 4 weeks before study drug administration;
4. Hepatocellular carcinoma confirmed by alpha-fetoprotein rate < 50 mg/dL no longer than 3 months before inclusion;
5. Signs of encephalopathy (grade 1 to 4 e.g. moderate to severe);
6. Presence of clinical ascites (slight to severe);
7. Drug addict patients treated with methadone or buprenorphine;
8. Presence of clinical ascites and/or pleural effusion. According to the investigator's judgement, small ascites radiologically detected but not clinically relevant could be accepted;
9. Severe hepatic encephalopathy, (Grade > 2, portal systemic encephalopathy score);
10. Recent history of gastrointestinal bleeding due to esophageal varices. According to the investigator's judgement, patient who had esophageal varices can be included if surgically treated by ligation, or sclerosis and with a prophylactic treatment by non-selective β-blockers (e.g., propranolol) and after checking by echography.
11. History of hepatic cytolysis due to medication;
12. Disorders or surgery of the gastrointestinal tract which may interfere with drug absorption or may otherwise influence the pharmacokinetics of the investigational medicinal product (e.g., inflammatory bowel disease, resections of the small or large intestine, etc.);
13. History of febrile illness within 5 days prior to dosing;
14. Any forbidden drug (as defined in protocol) intake during the 2 weeks or 5 half-lives of the drug preceding the first administration.

For Healthy Subjects with normal hepatic function:

1. Any history or presence of cardiovascular, pulmonary, gastro-intestinal, hepatic, renal, metabolic, hematological, neurologic, psychiatric, systemic, infectious or allergic disease
2. Frequent headaches (> twice a month) and / or migraines, recurrent nausea and / or vomiting;
3. Symptomatic hypotension whatever the decrease of blood pressure or asymptomatic postural hypotension defined by a decrease in SBP or DBP equal to or greater than 20 mmHg within two minutes when changing from the supine to the standing position;
4. Inability to abstain from intensive muscular effort;
5. History or presence of alcohol abuse (alcohol consumption > 40 grams/day);
6. Any drug intake (except paracetamol 3g/d) during the 2 weeks or 5 half-lives of the drug preceding the first administration;
7. Subject who would receive more than 4500 euros as indemnities for his participation in biomedical research within the 12 last months, including the indemnities for the present study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 15 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
Area under curve from dosing time to last measurment (AUC (0-t)) for MD1003 | predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  Blood samples will be collected
Area under curve from dosing tme to infinity (AUC(0-∞)) for MD1003 | predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  Blood samples will be collected
Observed maximum plasma concentration (Cmax) for MD1003 | predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  Blood samples will be collected
Measurement of concentration of MD1003 | predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  Blood samples will be collected
Measurement of concentration of Bisnorbiotin | predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  Blood samples will be collected
Measurement of concentration of Biotin sulfoxide | predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  Blood samples will be collected

SECONDARY OUTCOMES:
Measurement of plasma elimination half-life (t1/2) for MD1003 | predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  Blood samples will be collected
Measurement of time to reach observed maximum plasma concentration (tmax) for MD1003 | predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  Blood samples will be collected
Measurement of apparent volume of distribution (Vd/F) for MD1003 | predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  Blood samples will be collected
Measurement of elimination rate constant (Kel) for MD1003 | predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  Blood samples will be collected
Measurement of percentage of extrapolated AUCinf (%AUCextra) for MD1003 | predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  Blood samples will be collected
Measurement of apparent clearance (CL/F) for MD1003 | predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  Blood samples will be collected
Area under curve from dosing time to last measurment (AUC (0-t)) for Bisnorbiotin | predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  Blood samples will be collected
Area under curve from dosing time to last measurment (AUC (0-t)) for Biotin sulfoxide | predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  Blood samples will be collected
Area under curve from dosing tme to infinity (AUC(0-∞)) for Bisnorbiotin | predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  Blood samples will be collected
Area under curve from dosing tme to infinity (AUC(0-∞)) for Biotin sulfoxide | predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  Blood samples will be collected
Observed maximum plasma concentration (Cmax) for Bisnorbiotin | predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  Blood samples will be collected
Observed maximum plasma concentration (Cmax) for Biotin sulfoxide | predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  Blood samples will be collected
Measurement of time to reach observed maximum plasma concentration (tmax) for Bisnorbiotin | predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  Blood samples will be collected
Measurement of time to reach observed maximum plasma concentration (tmax) for Biotin sulfoxide | predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  Blood samples will be collected
Measurement of plasma elimination half-life (t1/2) Bisnorbiotin | predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  Blood samples will be collected
Measurement of plasma elimination half-life (t1/2) Biotin sulfoxide | predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  Blood samples will be collected
Measurement of elimination rate constant (Kel) for Bisnorbiotin | predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  Blood samples will be collected
Measurement of elimination rate constant (Kel) for Biotin sulfoxide | predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  Blood samples will be collected
Measurement of percentage of extrapolated AUCinf (%AUCextra) for Bisnorbiotin | predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  Blood samples will be collected
Measurement of percentage of extrapolated AUCinf (%AUCextra) for Biotin sulfoxide | predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  Blood samples will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Yves Donazzolo, MD, Principal Investigator — Eurofins Optimed
Locations (3):
- Eurofins Optimed, Gières, France
- Hungary (2):
  - DRC Drug Research Center Ltd., Balatonfüred
  - Clinical Research Units Hungary Ltd., Miskolc